CLINICAL TRIAL: NCT02319694
Title: Intraoperative Analysis of Reward and Impulsivity in the Basal Ganglia
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Other Study IDs: Pro00045557; R21NS084176 (NIH)
Record Dates: First submitted 2014-12-15; First posted 2014-12-18 (Estimated); Last update posted 2018-06-01 (Actual); Status verified 2018-05

CONDITIONS: Parkinson's Disease
Keywords: Basal Ganglia; Behavior; Behavioral; Brain; Cognitive; Computer Simulation; Cues; Data; Deep Brain Stimulation; Disease
MeSH Terms: conditions — Parkinson Disease; Behavior; Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No

SUMMARY:
This project studies the impulsive side effects of common treatments for Parkinson's Disease. By learning how parts of the brain involved in Parkinson's encode information related to reward and motivation, the investigators will better understand the reasons why Parkinson's patients often suffer from compulsive gambling, hypersexuality, and repetitive tinkering ("punding"). These results may lead to the design of better methods of deep brain stimulation (DBS) that minimize the behavioral side effects of Parkinson's treatment.

DETAILED DESCRIPTION:
While the typical treatments for Parkinson's disease (PD), dopaminergic drugs and deep brain stimulation (DBS), are proven to be effective in mitigating the motor deficits associated with the disease, these same methods also give rise to behavioral side effects including compulsive gambling, hypersexuality, and complex, purposeless stereotyped behavior ("punding"). And while much work has investigated the underlying patterns of neural activity giving rise to tremor, rigidity, and other motor effects of D, little is known about the neural genesis of impulsive side effects in humans. The investigators propose to characterize the patterns of neural activity underlying these failures of impulse control in an actual PD patient population undergoing surgery for the implantation of DBS electrodes. Such procedures offer a unique opportunity to collect data at the single neuron level in humans, since surgeons rely on intraoperative electrophysiology to identify the anatomical boundaries of the subthalamic nucleus (STN), the typical target of DBS in PD. Using multi-channel Ad-Tech microwire arrays, the investigators will simultaneously record multiple channels of single unit activity (both spikes and field potentials ) in STN and nearby structures while subjects perform cognitive tasks with validated links to impulsivity in human populations. In the balloon analogue risk task (BART) participants must balance risk and reward as they decide when to stop inflating a computerized balloon whose point value and risk of popping both grow with size. In the stop signal reaction task (SSRT), participants must respond as quickly as possible when a "go" cue appears, but countermand this response when a "stop" tone is played. At the neural level, the BART allows us to elucidate correlates of risk, outcome (both rewarding and aversive), and anticipation, while the SSRT, a well-studied model of impulsivity in both animal models and humans with strong links to computational models, will allow us to determine not only single unit but network-level patterns of activity underlying failures in impulse control. Through these experiments, as well as computational modeling, the investigators will characterize neural correlates of impulsivity in PD patients that will allow for the design of DBS protocols that mitigate impulsive side effects. The R21 mechanism will be used to further develop and streamline the process of multichannel recording and cognitive testing in the intraoperative setting and validate the hypothesized link between single neuron activity and models of behavior in the stop signal task.

ELIGIBILITY:
Inclusion Criteria:

* scheduled for implantation of deep brain stimulation device
* appropriate for awake surgery
* interest in participation

Exclusion Criteria:

* none

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants are patients scheduled to be implanted with Deep Brain Stimulation devices for treatment of Parkinson's Disease or Essential Tremor.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2013-07; Primary Completion 2017-02-27 (Actual); Study Completion 2017-02-27 (Actual)

PRIMARY OUTCOMES:
Brain activity data | during treatment
  Extracellular voltage measurements (microelectrode recording) from single and multi-neuron activity in the basal ganglia.
  Local field potentials from the same recording sites.
Behavioral data | during treatment
  Interactions of patients with a video game task, including joystick button responses, points earned, and response times.